Study Title: Veterans' perspectives on emergency room based lethal means safety interventions

**Principal Investigator:** REDACTED

**COMIRB No:** 20-2859 **Version Date:** 01.05.22

You are being asked to be in this research study because you are a Veteran who recently received care in the Emergency Department or Urgent Care.

If you join the study, you will be asked to speak with study staff by telephone or videoconference software. This overall research study is expected to take approximately 4 months. Your individual participation in the project will last approximately 2 hours.

This study is designed to learn more about how Veterans manage their access to household or personal medications and firearms.

Possible discomforts or risks include being asked to answer questions that make you feel uncomfortable or upset. You may feel frustrated or tired while completing the questionnaires. If this happens, you may pause or stop the study. You can also decline to answer any questions you do not feel comfortable answering. You may also call the Veteran's Crisis Line, emergency services, or the study team if you have significant concerns at any point during this study. We will do all we can to protect your information, but it cannot be guaranteed. There may be other risks the researchers have not thought of.

This study is not designed to benefit you directly.

Every effort will be made to protect your privacy and confidentiality by storing records about you in password protected or user-restricted files protected by the VA electronic security systems. Only members of the research team will have access to these data.

Some things we cannot keep private. If you indicate that you are going to physically hurt yourself, we have to report that to your mental health provider or emergency services. If you indicate you are going to physically hurt someone else, we have to report this to local authorities, command, and/or your mental health provider. If we get a court order to turn over your study records, we will have to follow the court order.

This research is being paid for by the U.S. Department of Veterans Affairs.

There is no cost to you for participation in this study. This research is being paid for by the VA Health Services Research and Development Service. You will be paid \$40, in the form of direct deposit or mailed check, for your participation. If you leave the study early or if we need to remove you from the study early, you will be paid \$20 per hour of your time, up to \$40. It is important to know that payments from participation in a study are taxable income. Your SSN will be collected and used to report this taxable income to the IRS.

The data we collect will be used for this study but may also be important for future research. Your data may be used for future research or distributed to other researchers for future study without additional consent if information that identifies you is removed from the data.

You have a choice about being in this study. You do not have to be in this study if you do not want to be. Taking part in this study is voluntary. You can choose to stop participating in this study at any time. You can also decline to answer any questions that you do not feel comfortable answering. If you refuse or decide to withdraw later, you will not lose any benefits or rights to which you are entitled.

Postcard Consent Template

CF-157, Effective 9-10-2018

If you have questions, you can call the study's Principal Investigator, REDACTED. You can call and ask questions at any time. You may have questions about your rights as someone in this study. If you have questions, you can call COMIRB (the responsible Institutional Review Board) at REDACTED. If you want to verify that this study is approved, please contact the VA Research Office at REDACTED.